CLINICAL TRIAL: NCT05905861
Title: Scalpel Versus Diathermy for Transverse Abdominal Incision in Women Undergoing First Elective Caesarean Section: a Randomized Controlled Trial
Brief Title: Scalpel Versus Diathermy for Transverse Abdominal Incision in First Elective Caesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Prof.Amerigo Vitagliano, MD, PhD, Assistant Professor (Researcher type-B), Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0049112
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Cesarean Section; Intraoperative Blood Loss; Postoperative Pain; Wound Heal
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group_A: skin incision with scalpel. (Placebo Comparator): In the scalpel group, the skin incision will be made using the traditional method, with a scalpel (No. 22).
  Interventions: Procedure: Skin incision with scalpel.
- Group_B: skin incision with diathermy. (Active Comparator): In the diathermy group, the incision will be made using a small flat blade pen electrode without applying pressure. The electrode will be set to cutting mode, delivering a sinusoidal current of maximum 120 watts.
  Interventions: Procedure: Skin incision with a diathermy.

INTERVENTIONS:
Procedure: Skin incision with scalpel. — A Pfannenstiel skin incision will be performed using a scalpel, extending through the subcutaneous tissue and rectus sheath. After separation of rectus muscles, peritoneum will be visualized and opened. Optimal hemostasis will be achieved by applying pressure to skin blood vessels and ligating any subcutaneous bleeding.
  Group A: skin incision with a scalpel.
  Arms: Group_A: skin incision with scalpel.
Procedure: Skin incision with a diathermy. — A Pfannenstiel skin incision will be made using a scalpel. Subsequently, a diathermy pen electrode will be employed for the dissection of deeper tissues.
  Optimal hemostasis will be achieved by using the same blade pen electrode, set to coagulation mode.
  Group B: skin incision with diathermy.
  Arms: Group_B: skin incision with diathermy.

SUMMARY:
The objective of this study will be to compare two methods of skin incisions during the first caesarean section (CS), that is scalpel and diathermy, assessing differences in blood loss during incision, incisional time, total surgery time, post-operative pain, wound healing, complications, and cosmetic outcomes.

DETAILED DESCRIPTION:
The scalpel has been historically used as the primary cutting tool during caesarean section (CS). However, advancements in surgical devices have introduced alternatives, such as the option to make a diathermic cut using electrosurgical units.

General surgeons have extensively demonstrated the advantages of diathermy over the scalpel for abdominal wall incisions, including faster opening time, reduced incisional blood loss, decreased post-operative pain, and a comparable wound complication rate.

In obstetrics, there is a scarcity of evidence in this regard, and no consensus or guidelines have been established regarding the optimal method for making a transverse abdominal incision during the first elective CS. Currently, the choice between using a scalpel or diathermy remains at discretion of the obstetric surgeon. The objective of this study will be to compare both methods of skin incisions during the first CS, assessing differences in blood loss during incision, incisional time, total surgery time, post-operative pain, wound healing, complications, and cosmetic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Women without a history of previous cesarean section or other abdominal surgery
2. Age greater then 18 years (only adult patients)
3. Body Mass Index (BMI) between 18.5 and 29.9 kg/m2
4. Gestational age greater then 37 weeks (at term pregnancies)
5. No contraindications to spinal anesthesia
6. Indication to elective CS: extra-obstetrical reasons, failure of medical induction of labor, breech fetal presentation
7. Informed consent

Exclusion Criteria:

1. Women refusing to participate in the study
2. Women undergoing urgency or emergency cesarean deliveries
3. Women with a history of previous cesarean section or abdominal surgery
4. Women with multifetal pregnancies
5. Necessity of general anesthesia
6. Use of anticoagulants
7. Patients needing a median longitudinal abdominal section
8. Patients with pacemakers
9. Allergy to cephalosporins
10. Any medical disorder that can affect wound healing as diabetes, hypertension, hepatic or renal diseases, chronic anemia, chronic skin conditions, congenital or acquired bleeding diathesis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incision blood loss | During surgery
  This will be calculated by weighing the gauze pre and postoperatively (1mg = 1ml) after complete hemostasis will be achieved.

SECONDARY OUTCOMES:
Incision time | During surgery
  We will compare incisional time by using a digital clock. The incisional time will be established as follows: when skin incision will be made, the surgeon will verbally announce "start ". Once the parietal peritoneum will be opened, the surgeon will announce "stop". The incision time will be calculated as the difference between "start" and "stop" times.
Total surgery time | During surgery
  Total surgery time will be the time between the start of the skin incision and the completion of the skin suture.
Post-operative pain assessed by VAS | During the first three days after surgery
  Post-operative pain will be evaluated for each participant at 1, 4, 8, 16, 24, 48, 72 hours postoperatively, by using the Visual Analog Scale (VAS). The VAS consists of a 10 cm long horizontal line with its extremes marked as 'no pain' (0) and 'worst pain imaginable' (10).
Wound complications | During the first month after surgery
  Will include edema, seroma, hematoma, dehiscence, and infection. The wound will be evaluated 24h and 72h after surgery, before patients discharge. Then, outpatient wound evaluation will be made 7 and 30 days after surgery.
Cosmetic wound evaluation assessed by POSAS | One month after surgery
  The cosmetic aspect of the wound will be evaluated outpatient 30 days after surgery by using the Patient and Observer Scar Assessment Scale (POSAS), that is a questionnaire that was developed to assess scar quality. It consists of two separate six-item scales (Observer Scale and Patient Scale), both of which are scored on a 10-point rating scale (1 = best result; 10 = worst result).

CONTACTS AND LOCATIONS:
Overall Officials: Amerigo Vitagliano, MD, PhD, Principal Investigator — "Aldo Moro" University of Bari
Locations (1):
- Azienda Ospedaliero-Universitaria "Consorziale Policlinico", Bari, Italy